CLINICAL TRIAL: NCT00601718
Title: A Phase I/II Study of Vorinostat Plus Rituximab, Ifosphamide, Carboplatin, and Etoposide for Patients With Relapsed or Refractory Lymphoid Malignancies or Untreated T- or Mantle Cell Lymphoma
Brief Title: Vorinostat, Rituximab, Ifosfamide, Carboplatin, and Etoposide in Treating Patients With Relapsed or Refractory Lymphoma or Previously Untreated T-Cell Non-Hodgkin Lymphoma or Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Gopal, Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSOC 2302; NCI-2010-00870 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2008-01-24; First posted 2008-01-28 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Mycosis Fungoides/Sezary Syndrome; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Mycosis Fungoides/Sezary Syndrome; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Vorinostat; Rituximab; Ifosfamide; indolepropanol phosphate; Carboplatin; Etoposide; Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor, monoclonal antibody, chemotherapy (Experimental): Patients receive vorinostat PO QD on days 1-5, ifosfamide IV continuously over 24 hours and carboplatin IV over 1 hour on day 4, and etoposide IV over 1 hour on days 3-5. Patients who are CD20+ also receive rituximab IV once on day 3, 4, or 5. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Biological: rituximab; Drug: ifosfamide; Drug: carboplatin; Drug: etoposide; Other: pharmacological study; Other: laboratory biomarker analysis; Genetic: gene expression analysis

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies
Genetic: gene expression analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of vorinostat when given together with rituximab, ifosfamide, carboplatin, and etoposide and to see how well they work in treating patients with relapsed or refractory lymphoma or previously untreated T-cell non-Hodgkin lymphoma or mantle cell lymphoma. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as ifosfamide, carboplatin, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving vorinostat together with rituximab and combination chemotherapy may kill more cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine maximally tolerated dose of vorinostat that can be combined with RICE chemotherapy in patients with relapsed lymphoid malignancies.

II. To determine the safety and toxicity of the above regimen. III. To gain a preliminary assessment of the efficacy of the above regimen. IV. To determine the ability to proceed to peripheral blood stem cell collection following the above regimens (the impact of above regimen on stem cell reserve).

V. To describe vorinostat concentration attained at or near the MTD. VI. To evaluate the change of histone acetylation patterns and pro-apoptotic proteins of primary target (tumor) and non-target peripheral blood mononuclear cells (PBMC) cells following high-dose HDAC inhibition.

VII. To describe the gene expression profile changes of tumor and non-tumor cells following high-dose HDAC inhibition.

OUTLINE: This is a phase I/II dose-escalation study of vorinostat.

Patients receive vorinostat orally (PO) once daily (QD) on days 1-5, ifosfamide IV continuously over 24 hours and carboplatin IV over 1 hour on day 4, and etoposide IV over 1 hour on days 3-5. Patients who are CD20+ also receive rituximab IV once on day 3, 4, or 5. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have relapsed or primary refractory lymphoid malignancy (including B-cell, T-cell, or Hodgkins disease), or untreated T-NHL or MCL
* Patients with other lymphomas that have not received any prior therapy and are not candidates for anthracycline-based therapies, are eligible with PI review and approval
* Revised European American classification (REAL), or World Health Organization (WHO) classification of patient's malignancies must be provided
* Patients must have measurable disease defined as lesions that can be accurately measured in two dimensions by computed tomography (CT), magnetic resonance imaging (MRI), medical photograph (skin or oral lesion), plain x-ray, or other conventional technique and a greatest transverse diameter of 1 cm or greater; or palpable lesions with both diameters >= 2 cm
* Patients must have a bone marrow aspirate and biopsy within 28 days of enrollment and no intervening anticancer therapy
* Patients must have a CT of chest, abdomen, and pelvis within 28 days of enrollment; patients with evidence of adenopathy in the neck must have a CT of neck
* Patients should not have evidence of active central nervous system lymphoma
* Electrocardiogram (EKG) must be free of any arrhythmias (excluding sinus arrhythmia or infrequent premature ventricular contractions)
* Patients must have a Southwest Oncology Group (SWOG) performance status of 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Serum creatinine < 1.5 mg/dl or creatinine clearance greater than 60/ ml per minute by the following formula (all tests must be performed within 28 days prior to registration)
* Total bilirubin < 1.5 times upper limit of normal, aspartate aminotransferase (AST) < 5 times upper limit of normal
* Patients must have a serum lactate dehydrogenase (LDH) performed within 14 days prior to registration
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines
* Patients must be anticipated to complete at least 2 cycles of chemotherapy
* Platelets >= 100,000/mm^3 (without transfusion)

Exclusion Criteria:

* Patients known to be human immunodeficiency virus (HIV) positive
* Pregnant or nursing women; men or women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients with other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, cervical cancer in situ, or other cancer from which the patient has been disease free for 5 years or greater, unless approved by the protocol Chair or Co-Chair
* Patients that are refractory (i.e. not responded or progressed within 6 months) to a carboplatin, cisplatin, ifosfamide, or etoposide-based regimen-based regimen
* Patients that have other medical conditions that would contraindicate treatment with aggressive chemotherapy (including active infection, uncontrolled hypertension, congestive heart failure, unstable angina pectoris, or myocardial infarction within the past 6 months, or uncontrolled arrhythmia)
* Patients with a history of impaired cardiac status (including history of severe coronary artery disease, cardiomyopathy, congestive heart failure or arrhythmia); if the patient's history is questionable, a measurement of left ventricular ejection fraction should be obtained within 42 days prior to registration; patients with left ventricular ejection fraction < 50% are not eligible
* Autologous or allogeneic transplantation within 12 months or radioimmunotherapy within 6 months of registration
* No concurrent treatment with valproic acid or on valproic acid within 2 weeks of study enrollment
* No prior treatment with histone deacetylase inhibitors
* No concurrent therapy for this malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Budde, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Puget Sound Oncology Consortium, Seattle, Washington, United States

REFERENCES:
- [Background] Budde LE, Zhang MM, Shustov AR, Pagel JM, Gooley TA, Oliveira GR, Chen TL, Knudsen NL, Roden JE, Kammerer BE, Frayo SL, Warr TA, Boyd TE, Press OW, Gopal AK. A phase I study of pulse high-dose vorinostat (V) plus rituximab (R), ifosphamide, carboplatin, and etoposide (ICE) in patients with relapsed lymphoma. Br J Haematol. 2013 Apr;161(2):183-91. doi: 10.1111/bjh.12230. Epub 2013 Jan 29. PMID 23356514

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor, Monoclonal Antibody, Chemotherapy
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor, Monoclonal Antibody, Chemotherapy
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 56 [23 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Vorinostat
Time Frame: 28 days post last dose of study drug
Measure: Number; unit: mg twice daily X 5 days
Arm/Group | Treatment (Enzyme Inhibitor, Monoclonal Antibody, Chemotherapy
Number analyzed (Participants) | 29
mg twice daily X 5 days | 500

2. Primary Outcome: Safety and Toxicity According to CTCAE v3.0
Description: Common dose limiting toxicities.
Time Frame: 3-5 weeks post end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor, Monoclonal Antibody, Chemotherapy
Number analyzed (Participants) | 29
Participants
  Infection | 2
  Hypokalemia | 2
  Transaminitis | 2
  Grade 3 related gastrointestinal toxicity | 9

3. Primary Outcome: Efficacy (Response Rate) of Vorinostat Combined With RICE Chemotherapy
Time Frame: 3-5 weeks post end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor, Monoclonal Antibody, Chemotherapy
Number analyzed (Participants) | 29
Participants | 19

4. Primary Outcome: Ability to Proceed to Peripheral Blood Stem Cell Collection Following Treatment
Time Frame: 1-3 weeks post end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor, Monoclonal Antibody, Chemotherapy
Number analyzed (Participants) | 21
Participants | 20

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor, Monoclonal Antibody, Chemotherapy
Serious Adverse Events (participants affected / at risk) | 10/29
Other Adverse Events (participants affected / at risk) | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor, Monoclonal Antibody, Chemotherapy (N=29)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Nausea/Vomiting (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hypotension (Vascular disorders) | 1
Allergic reaction (Immune system disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor, Monoclonal Antibody, Chemotherapy (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Infection (Infections and infestations) | 8
Nausea (Gastrointestinal disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Hypophasphataemia (Metabolism and nutrition disorders) | 12
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 4
AST/ALT (Investigations) | 4
DVT (General disorders) | 2
Elevated PTT (General disorders) | 3
Pain (General disorders) | 4
Fatigue (General disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes